CLINICAL TRIAL: NCT06933628
Title: A Randomized Comparative Study of Customized Titanium Plates Versus Three-Dimensional (3D)-Printed Splints for Maxillary Repositioning Accuracy in LeFort I Orthognathic Surgery
Brief Title: Custom Titanium Plates vs. 3D Splints in LeFort I Osteotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Abdalkareem Mansour, Assistant Lecturer, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 887/1849
Record Dates: First submitted 2025-04-11; First posted 2025-04-18 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Dentofacial Deformities
Keywords: dentofacial deformities; customized titanium plates; PSI; virtual surgical planning; 3D printed splints
MeSH Terms: conditions — Dentofacial Deformities

STUDY DESIGN:
Intervention Model Description: Group I (Experimental Group): Patients whose surgery was guided by personalized orthognathic surgical guides. The maxillary segments were fixed using customized titanium plates designed through virtual surgical planning (VSP).
  Group II (Control Group): Patients whose surgery was guided by an intermediate splint designed based on the final virtual model and fabricated using computer-aided manufacturing (CAM) technology. Fixation was completed with conventional titanium miniplates and screws.
Who Masked: Participant, Outcomes Assessor
Masking Description: "Both the participants and outcome assessors were blinded to the method of virtual surgical planning (VSP) implementation-whether using customized titanium plates or 3D-printed splints-to minimize bias."
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- customized titanium plates group (Experimental): "Patients whose surgery was guided by a personalized orthognathic surgical guide, with the maxillary segments fixed using a pair of customized titanium plates."
  Interventions: Procedure: Patient-Specific Titanium Plates
- 3D printed splint group (Active Comparator): "Patients whose surgery was guided by an intermediate splint, designed based on the final virtual model and fabricated using computer-aided manufacturing (CAM) technology.
  Interventions: Procedure: 3D-Printed Intermediate Splint

INTERVENTIONS:
Procedure: Patient-Specific Titanium Plates — Custom 3D-printed titanium fixation plates and cutting guides
  Arms: customized titanium plates group
Procedure: 3D-Printed Intermediate Splint — CAD/CAM-fabricated occlusal splint for maxillary positioning
  Arms: 3D printed splint group

SUMMARY:
This randomized comparative study evaluates the accuracy and feasibility of two techniques for maxillary repositioning in Le Fort I osteotomy:

Customized titanium plates (splintless technique)

Three-dimensional (3D)-printed intermediate splints

Participants (n = 12) aged 18-30 years with dentofacial deformities will be equally divided into two groups:

Group I: Osteotomy guided by patient-specific surgical guides, fixed with pre-bent customized titanium plates.

Group II: Osteotomy guided by 3D-printed intermediate splints with conventional fixation.

Primary Outcome Accuracy of maxillary repositioning (measured as millimeter [mm] deviation from the virtual surgical plan), assessed via computed tomography (CT) superimposition using Mimics software at one week postoperatively.

Secondary Outcomes

Operative time

Fabrication accuracy of the customized titanium plate and 3D-printed splint

Postoperative complications (e.g., infection, plate failure)

Hypothesis Customized titanium plates will reduce maxillary positioning errors and operative time compared to 3D-printed splints.

Relevance This study may validate splintless techniques for improved precision in orthognathic surgery.

DETAILED DESCRIPTION:
Background and Rationale Orthognathic surgery relies on precise maxillary repositioning to achieve both functional and aesthetic outcomes. Traditional techniques using three-dimensional (3D)-printed splints are limited by potential errors in splint seating, condylar positioning, and vertical dimension control. Emerging splintless approaches using customized titanium plates and cutting guides-designed through virtual surgical planning (VSP)-may improve accuracy by eliminating interocclusal splints, preventing condylar sagging, and reducing operative time. This study compares these two techniques in Le Fort I osteotomy, addressing the evidence gap for splintless feasibility, particularly in resource-limited settings.

Study Design Type: Prospective, randomized, single-blind, parallel-group comparative trial.

Setting: Al-Azhar University, Faculty of Dental Medicine, and Sayyed Galal University Hospital (Cairo, Egypt).

Aim of the Study To assess the accuracy and stability of customized titanium plates versus the 3D-printed splint technique in Le Fort I osteotomy for orthognathic surgery.

Population Twelve patients (aged 18-30 years) with dentofacial deformities classified as American Society of Anesthesiologists (ASA) Class I or II, who do not require a segmental Le Fort I osteotomy, are not pregnant or suspected of pregnancy, and have no prior orthognathic surgery or facial anomalies.

Participants were randomized 1:1 into:

Group I (Experimental): Patient-specific cutting guides + customized titanium plates (splintless technique).

Group II (Comparator): 3D-printed intermediate splints + conventional fixation with miniplates and screws.

Blinding: Outcome assessors analyzing computed tomography (CT) scans was blinded to group allocation.

Interventions Preoperative Planning All patients underwent CT imaging (1 mm slices) and dental cast scanning using intraoral scanners to create stereolithography (STL) files. The composite model was merged using Mimics 21.0 software for virtual surgical planning (VSP). Orthopantomography was used to evaluate dentition. Lateral cephalometry was performed for analytical planning.

Virtual Planning Process:

Occlusal registration

STL file production

Digital Imaging and Communications in Medicine (DICOM) file generation

Surgical simulation

Transfer method planning

Digital dental models were generated via high-resolution scanning and merged with the 3D skull model to replace the less accurate CT dental data, resulting in a highly accurate composite skull model using Mimics Medical 21.0 (Materialise NV, Leuven, Belgium).

Group I: The customized titanium plate system included a pair of cutting guides with preplanned screw holes and a pair of custom fixation plates. STL files were exported for fabrication using two 3D printers.

Group II: Teeth-borne 3D intermediate splints were designed and printed to guide surgical movement of osteotomized segments.

Surgical Procedures All patients were admitted to the hospital and underwent routine lab investigations and specialty evaluations (cardiac, thoracic, internal medicine). Surgery was performed under general anesthesia with sterile preparation.

Le Fort I Osteotomy:

A standard Le Fort I osteotomy was performed via a maxillary vestibular approach (incision from upper first molar to opposite first molar, 5 mm above the mucogingival junction).

The flap was elevated to fit the cutting guide. Osteotomies were performed on the lateral maxillary wall, lateral nasal wall, nasal septum, and pterygoid plates. The maxilla was disimpacted and repositioned:

Group I: Fixed using customized titanium plates.

Group II: Repositioned using a 3D-printed splint and fixed with conventional titanium miniplates.

Bilateral Sagittal Split Osteotomy (BSSO):

Performed through the mandibular vestibular approach.

The incision extended from the anterior border of the ramus to the lower first molar.

Osteotomy began at the medial ramus wall above the mandibular foramen, extended to the anterior border, and completed with a vertical cut to the mandible's lower border.

Mandibular segments were repositioned with intermediate splints in both groups. Surgery was only performed if indicated.

Group I (Splintless):

Maxillary cutting guides were fixed in position based on unique anatomical features of the maxillozygomatic buttress and anterior wall.

Cutting lines and screw holes were marked.

After removing the guides, osteotomies were completed, and the maxilla was repositioned and fixed with custom titanium plates and screws.

Group II (3D-Printed Splint):

Osteotomized jaw segments were aligned using the 3D-printed intermediate splint.

Intermaxillary fixation was applied, followed by rigid fixation with conventional miniplates and screws.

Postoperative Protocol CT scans were performed one week postoperatively to assess accuracy of cutting guides, customized titanium plates, and 3D-printed splints.

Follow-up: Clinical evaluations at 1 week, 1 month, 3 months, 6 months, and 12 months to assess occlusion and complications.

Outcomes Primary outcome: Maxillary repositioning accuracy (mm deviation from VSP) CT superimposition (Mimics 21.0)

Secondary outcomes:

Operative time (incision-to-fixation)

Fabrication accuracy of customized plate and 3Dprinted splint:

* Outcome occlusion (Canine/Angle classification)
* Complication rates (infection, plate failure, sensory deficits) Clinical records Statistical Analysis Sample Size: n = 6 per group (80% power, α = 0.05, effect size d = 1.94-2.18), based on Karanxha et al. (2020).

Tests:

Independent t-tests or Mann-Whitney U tests for intergroup comparisons. Paired t-tests for pre- vs. postoperative CT deviations. Software: SPSS v26 Significance threshold: p < 0.05

Ethical and Regulatory Considerations IRB Approval: Granted by Al-Azhar University (protocol attached).

Informed Consent: Written informed consent obtained from all participants (Arabic language).

Data Handling: All CT data and models anonymized and securely stored. Only aggregated results will be published.

ELIGIBILITY:
Inclusion Criteria:

Patients with dentofacial deformities requiring Le Fort I orthognathic surgery. Patients aged between 18 and 30 years. Medically healthy patients classified as American Society of Anesthesiologists (ASA) Class I or II.

Exclusion Criteria:

Patients requiring a segmental Le Fort I osteotomy. Patients with suspected or confirmed pregnancy. Patients with a previous history of orthognathic surgery. Patients with cleft palate or other craniofacial anomalies.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Accuracy of custom-made plate vs 3D printed splint | postoperative one week
  Accuracy of Outcomes of Custom-Made Plate and 3D-Printed Splint The accuracy of outcomes for both the custom-made titanium plates and the 3D-printed splints will be assessed by comparing the planned virtual outcomes to the actual postoperative results. Postoperative computed tomography (CT) scans will be superimposed onto the planned models using the Mimics Medical 21.0 software (Materialise NV, Leuven, Belgium). The discrepancies between the planned and actual outcomes will be measured in millimeters to evaluate surgical accuracy.

CONTACTS AND LOCATIONS:
Overall Officials: wael A El-Mohandes, professor, Study Chair — Al-Azhar University
Locations (1):
- Sayyed Galal hospital, Cairo, Bab Al Sheraya. ELObera, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heufelder M, Wilde F, Pietzka S, Mascha F, Winter K, Schramm A, Rana M. Clinical accuracy of waferless maxillary positioning using customized surgical guides and patient specific osteosynthesis in bimaxillary orthognathic surgery. J Craniomaxillofac Surg. 2017 Sep;45(9):1578-1585. doi: 10.1016/j.jcms.2017.06.027. Epub 2017 Jul 8. PMID 28793965
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/28793965/